CLINICAL TRIAL: NCT01540058
Title: A Randomised Phase III Trial Comparing a Strategy Based on Molecular Analysis to the Empiric Strategy in Patients With Carcinoma of an Unknown Primary (CUP)
Brief Title: Trial Comparing a Strategy Based on Molecular Analysis to the Empiric Strategy in Patients With CUP
Acronym: GEFCAPI04
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2011-A01202-39; 2011/1751 (Other: CSET number)
Record Dates: First submitted 2012-02-13; First posted 2012-02-28 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Neoplasms, Unknown Primary
MeSH Terms: conditions — Neoplasms, Unknown Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- test-guided strategy (Experimental): Treatment considered as the standard at the time of patient inclusion based on the primary cancer suspected by "the BioTheranostics Cancer Type ID test" molecular analysis
  Interventions: Other: Cancer Type ID test
- Empiric strategy (Active Comparator): Gemcitabine/Cisplatin
  Interventions: Other: No test Empiric strategy

INTERVENTIONS:
Other: Cancer Type ID test — CancerTYPE ID is a real-time RT-PCR assay that measures and interprets the differential expression of 92 genes as a molecular correlate for tumor classification. The test classifies 28 main tumor types and 50 subtypes using an algorithm incorporating gene expression data from a reference database of 2,094 tumor specimens. CancerTYPE ID is used, in conjunction with other clinical and diagnostic procedures, to help identify tumor type and histological subtype. The performance characteristics and reproducibility of the test have been published previously (Erlander et al., 2011 ; Kerr et al., 2012).
  CancerTYPE ID is conducted on formalin-fixed paraffin-embedded (FFPE) tumor specimens at bioTheranostics' high complexity laboratory, which is certified by Clinical Laboratory Improvement Amendments (CLIA), accredited by the College of American Pathologists (CAP), and approved by the State of New York.
  Arms: test-guided strategy
Other: No test Empiric strategy — Empiric strategy
  Arms: Empiric strategy

SUMMARY:
This is a european randomised, phase III, multi-centric study comparing a diagnostic and therapeutic strategy based on molecular analysis followed by suspected primary cancer tailored specific therapy, to an empiric strategy in patients with carcinoma of unknown primary. The purpose of this trial is to determine whether or not a strategy based on molecular analysis is effective in improving the progression free survival rates of patients with carcinoma of unknown primary (CUP).

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with carcinoma of unknown primary, confirmed by histopathological analysis (including an immunohistochemical analysis) and corresponding to one of the following histologic types : moderately or well-differentiated adenocarcinoma, poorly-differentiated adenocarcinoma, undifferentiated carcinoma, squamous-cell carcinoma
2. Diagnostic work-up in keeping with Standard Options Recommandations des CAPI (Lesimple et al., 2003),
3. Age > 18 years,
4. Performance Status 0, 1 or 2 according to ECOG
5. Good or poor prognosis CUP classified according to the GEFCAPI classification
6. CUP with at least one measurable lesion
7. Tumour sample available for molecular analysis
8. CUP not belonging to a subgroup requiring a specific treatment,
9. Satisfactory haematological, renal and hepatic function
10. Cardiac, respiratory and neurological function compatible with the administration of cisplatin chemotherapy,
11. No previous chemotherapy for a CUP
12. Previous radiotherapy is acceptable, but it should be completed at least 4 weeks before the start of systemic treatment. Randomization can be performed during this time frame.
13. All patients with reproductive potential must practice an effective method of birth control throughout the study. Female patients with childbearing potential must have a negative pregnancy test within 7 days before study treatment
14. Information delivered to patient and informed consent form signed by the patient or legal representative.

Exclusion Criteria:

1. Patients in whom the diagnosis has not been histologically confirmed (a cytological analysis alone does not permit patient entry onto the trial),
2. Patients with known HIV infection
3. Patients with symptomatic brain metastases,
4. Associated disease likely to prevent the patient from receiving the treatment,
5. Previous history of cancer (excepted skin basocellular epithelioma or epithelioma in situ of the uterine cervix) during the 5 years before study entry,
6. Patients already included in another clinical trial with an experimental therapy,
7. Pregnant woman or woman who are breastfeeding,
8. Compliance with trial medical follow-up impossible due to geographic, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2012-03-22 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first progression or date of death from any cause, whichever came first, assessed up to 18 months
  Progression according to RECIST criteria or death of any cause.

SECONDARY OUTCOMES:
Response rate | An expected average of 1 year
  Response will be assessed using RECIST criteria
Tolerance (Toxicity grade III and IV, toxic death) | An expected average of 1 year
  Toxicity will be assessed using NCI-CTC criteria version 4.0
Overall survival | From the day of randomization to death or last date of follow-up, assessed up to 18 months
  Death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Karim FIZAZI, MD, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (3):
- Rigshospitalet, Copenhagen, Denmark
- Institut Gustave Roussy, Villejuif, Val De Marne, France
- Viecuri Medical Centre Venlo, Venlo, Netherlands